CLINICAL TRIAL: NCT03923699
Title: Telemedicine Control Tower for the Operating Room: Navigating Information, Care and Safety - Randomized Pragmatic Trial
Brief Title: Telemedicine Control Tower for the Operating Room: Navigating Information, Care and Safety
Acronym: TECTONICS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201903026; R01NR017916 (NIH)
Record Dates: First submitted 2019-03-06; First posted 2019-04-23 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Surgery; Surgery--Complications; Perioperative/Postoperative Complications
Keywords: Telemedicine; Anesthesia Control Tower; Machine Learning; Forecasting Algorithms; Decision Support; Randomized Controlled Trial
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Randomized Parallel assignment
Who Masked: Participant
Masking Description: Anesthesia practitioner un-blinded to intervention, subject blinded to intervention, data analyst blinded to intervention, ACT Clinicians un-blinded to intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of care arm (No Intervention): Operating rooms in the standard of care group will be monitored but, the ACT clinicians will not contact the operating room unless it is clinically necessary for patient safety purposes.
- Anesthesia Control Tower monitoring (Experimental): Clinicians in the Anesthesiology Control Tower will provide extra support for the anesthesiology team in the operating room using AlertWatch and integrating machine-learning forecasting algorithms for adverse outcomes.
  Interventions: Device: Anesthesia Control Tower monitoring

INTERVENTIONS:
Device: Anesthesia Control Tower monitoring — Real time data will be monitored through the AlertWatch® system as well as the patient's EHR.
  Arms: Anesthesia Control Tower monitoring

SUMMARY:
Medical errors account for thousands of potentially preventable deaths each year. With the annual increase of surgical cases there is a need for research into the potential utility of a telemedicine-based control center for the operating room to assess risk, diagnose negative patient trajectories, implement evidence-based practices, and improve outcomes.

DETAILED DESCRIPTION:
This will be a single center, randomized, controlled, phase 3 pragmatic clinical trial. Forty-eight operating rooms will be randomized daily to receive support from the ACT or not. All adults (eighteen years and older) undergoing surgical procedures in these operating rooms will be included and followed until 30-days after their surgery. Clinicians in operating rooms randomized to 'intervention' will receive decision support from clinicians in the ACT. In operating rooms not randomized to receive decision support from the ACT, the current standard of anesthesia care will be delivered. The intention-to-treat principle will be followed for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years or older undergoing surgery at Barnes Jewish Hospital in St. Louis, MO

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79560 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Avidan, MBBCh, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers as the data is collected under a waiver of informed consent and is also protected by a Certificate of Confidentiality from the NIH.

REFERENCES:
- [Derived] King CR, Fritz BA, Gregory SH, Budelier TP, Ben Abdallah A, Kronzer A, Helsten DL, Torres B, McKinnon SL, Tripathi S, Abdelhack M, Goswami S, Montes de Oca A, Mehta D, Valdez MA, Karanikolas E, Higo O, Kerby P, Henrichs B, Wildes TS, Politi MC, Abraham J, Avidan MS, Kannampallil T; ACTFAST collaborator group. Effect of telemedicine support for intraoperative anaesthesia care on postoperative outcomes: the TECTONICS randomised clinical trial. Br J Anaesth. 2025 Mar;134(3):671-680. doi: 10.1016/j.bja.2024.11.017. Epub 2025 Jan 3. PMID 39753404
- [Derived] King CR, Fritz BA, Gregory SH, Budelier TP, Ben Abdallah A, Kronzer A, Helsten DL, Torres B, McKinnon SL, Tripathi S, Abdelhack M, Goswami S, de Oca AM, Mehta D, Valdez MA, Karanikolas E, Higo O, Kerby P, Henrichs B, Wildes TS, Politi MC, Abraham J, Avidan MS, Kannampallil T; ACTFAST collaborator group. Effect of Telemedicine Support for Intraoperative Anaesthesia Care on Postoperative Outcomes: The TECTONICS Randomised Clinical Trial. medRxiv [Preprint]. 2024 Nov 26:2024.05.21.24307593. doi: 10.1101/2024.05.21.24307593. PMID 38826207
- [Derived] Fritz B, King C, Chen Y, Kronzer A, Abraham J, Ben Abdallah A, Kannampallil T, Budelier T, Montes de Oca A, McKinnon S, Tellor Pennington B, Wildes T, Avidan M. Protocol for the perioperative outcome risk assessment with computer learning enhancement (Periop ORACLE) randomized study. F1000Res. 2022 Sep 29;11:653. doi: 10.12688/f1000research.122286.2. eCollection 2022. PMID 37547785
- [Derived] King CR, Abraham J, Kannampallil TG, Fritz BA, Ben Abdallah A, Chen Y, Henrichs B, Politi M, Torres BA, Mickle A, Budelier TP, McKinnon S, Gregory S, Kheterpal S, Wildes T, Avidan MS; TECTONICS Research Group. Protocol for the Effectiveness of an Anesthesiology Control Tower System in Improving Perioperative Quality Metrics and Clinical Outcomes: the TECTONICS randomized, pragmatic trial. F1000Res. 2019 Nov 29;8:2032. doi: 10.12688/f1000research.21016.1. eCollection 2019. PMID 32201572

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Operating Room Days
Period: Overall Study
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Started | 39750; 17907 Operating Room Days | 39810; 18091 Operating Room Days
Completed | 39750; 17907 Operating Room Days | 39810; 18091 Operating Room Days
Not Completed | 0; 0 Operating Room Days | 0; 0 Operating Room Days

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring | Total
Number analyzed (Participants) | 39750 | 39810 | 79560
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (17.0) | 57.2 (16.8) | 57.2 (16.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 19752 | 19813 | 39565
  Male | 19994 | 19992 | 39986
  Unknown or Other | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 112 | 111 | 223
  Asian | 417 | 453 | 870
  Native Hawaiian or Other Pacific Islander | 58 | 63 | 121
  Black or African American | 7776 | 7875 | 15651
  White | 27595 | 27628 | 55223
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3792 | 3680 | 7472
Region of Enrollment [Number; unit: participants]
  United States | 39750 | 39810 | 79560
ASA Physical Status [Count of Participants; unit: Participants] — Range, 1 to 6; 1 indicates healthy, 2 indicates mild systemic disease, 3 indicates severe systemic disease, 4 indicates severe systemic disease that is a constant threat to life, 5 indicates not expected to survive without surgery, 6 indicates neurologically deceased organ donor. In this study, only patients with an ASA 1 to 5 were collected.
  Participants
    ASA 1 | 1406 | 1413 | 2819
    ASA 2 | 12071 | 12117 | 24188
    ASA 3 | 17295 | 17282 | 34577
    ASA 4 | 4009 | 4034 | 8043
    ASA 5 | 132 | 120 | 252
    Unknown or Other | 4837 | 4844 | 9681

OUTCOME MEASURES:

1. Primary Outcome: Thirty-day Postoperative Mortality
Description: This will include death of any cause occurring in or out of the hospital, within 30 days of the index surgery.
Time Frame: 30 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 39750 | 39810
Participants | 899 | 866
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.41, Regression, Poisson — Not adjusted for multiple comparisons; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.85 to 1.08]

2. Primary Outcome: Number of Participants With Postoperative Delirium
Description: Defined as an acute change in consciousness or cognition. It has a fluctuating course, and is characterized by inattention, disorganized thinking and altered level of consciousness. The institution has trained the nursing staff on our surgical intensive care units to assess all patients for postoperative delirium using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) instrument.
Time Frame: 7 days post-op
Population: Patients that did not have a CAM-ICU performed, or CAM-ICU scores within 30 minutes of a documented deep level of sedation (Richmond Agitation Sedation Scale < -3) are excluded. All other delirium assessments within 7 days will be included, with any positive evaluations yielding a positive event.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 4711 | 4681
Participants | 1506 | 1502
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.92, Regression, Poisson — Not adjusted for multiple comparisons; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.92 to 1.10]

3. Primary Outcome: Number of Participants With Postoperative Respiratory Failure
Description: Defined as mechanical ventilation for greater than 24 hours after surgery, or unplanned postoperative re-intubation and mechanical ventilation within 30 days of surgery.
Time Frame: 30 days post-op
Population: Patients with tracheostomies and preoperative ventilation are excluded. Airway events within 24 hours after surgeries within 30 days of the index operation are excluded. That is, a 24 hour window of ventilation is allowed after all surgeries without triggering a positive event.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 37600 | 37652
Participants | 1301 | 1282
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.68, Regression, Poisson — Not adjusted for multiple comparisons; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.89 to 1.09]

4. Primary Outcome: Number of Participants With Postoperative Acute Kidney Injury
Description: Diagnosed when any of the following three criteria are met: (i) an increase in serum creatinine by 50% compared with preoperative within 7 days, (ii) any increase in serum creatinine > 0.3 mg/dL in 48 hours, or (iii) oliguria (urine output <0.5 mL/kg/hr for 6-12 hours).
Time Frame: 7 days post-op
Population: Patients with diagnosed renal failure, serum creatinine >4 mg/dl, and dialysis in the last week are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 37240 | 37393
Participants | 2784 | 2736
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.42, Regression, Poisson — Not adjusted for multiple comparisons; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.92 to 1.05]

5. Secondary Outcome: Temperature Management
Description: Percentage of patients with Temperature ≥ 36°C at end of surgery.
Time Frame: 1 day
Population: Patients with missing secondary outcomes are not included in the analysis of those outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 34340 | 34711
Participants | 27101 | 27398
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.99, Regression, Poisson — Not adjusted for multiple comparisons; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.98 to 1.02]

6. Secondary Outcome: Antibiotic Redosing
Description: Percentage of patients with antibiotic redosing compliant with guidelines developed by the institutional pharmacy and therapeutics committee.
Time Frame: 1 day
Population: Patients without an indicated redosing event are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 5811 | 5919
Participants | 5520 | 5629
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.95, Regression, Poisson — Not adjusted for multiple comparisons; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.95 to 1.05]

7. Secondary Outcome: Mean Arterial Pressure Management
Description: Percentage time during surgery with mean arterial pressure ≥ 60 mmHg
Time Frame: 1 day
Population: Patients with missing secondary outcomes are not included in the analysis of those outcomes.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 39032 | 39127
percentage of time | 0.96 (0.08) | 0.96 (0.08)
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.29, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.00 to 0.00]

8. Secondary Outcome: Mean Airway Pressure With Mechanical Ventilation
Description: Percentage time during surgery with low PIP (peak inspiratory pressure)
Time Frame: 1 day
Population: Patients with missing secondary outcomes are not included in the analysis of those outcomes.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 30306 | 30573
percentage of time | 0.92 (0.21) | 0.92 (0.22)
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.37, Regression, Linear — Not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.01 to 0.00]

9. Secondary Outcome: Blood Glucose Management
Description: Percentage of patients with blood glucose ≥ 200 mg/dL at end of surgery.
Time Frame: 1 day
Population: Patients with missing secondary outcomes are not included in the analysis of those outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 32435 | 32437
Participants | 1786 | 1848
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.30, Regression, Poisson — Not adjusted for multiple comparisons; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.95 to 1.13]

10. Secondary Outcome: Measured Anesthetic Concentration
Description: Percentage of patients without ≥ 15 consecutive min of anesthetic concentration ≤ 0.3 MAC during anesthetic maintenance period.
Time Frame: 1 day
Population: Patients with doses of sedatives at greater than the following dose-rates are excluded: Propofol > 40 mcg/kg/min, Ketamine > 0.3 mg/kg/hr. Patients with missing secondary outcomes are not included in the analysis of those outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 30175 | 30460
Participants | 29851 | 30087
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.85, Regression, Poisson — Not adjusted for multiple comparisons; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.98 to 1.02]

11. Secondary Outcome: Fresh Gas Flow Rates
Description: Percentage of patients with efficient fresh gas flow for ≥90% of the anesthetic maintenance period.
Time Frame: 1 day
Population: Only times with > 0.3 age adjusted MAC are included. Patients with missing secondary outcomes are not included in the analysis of those outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
Number analyzed (Participants) | 26739 | 26837
Participants | 19899 | 19839
Statistical Analysis 1: Comparison: Standard of Care Arm vs Anesthesia Control Tower Monitoring; Test type: Superiority; p = 0.51, Regression, poisson — Not adjusted for multiple comparisons; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.97 to 1.02]

ADVERSE EVENTS:
Time Frame: 30 days post-op
Arm/Group | Standard of Care Arm | Anesthesia Control Tower Monitoring
All-Cause Mortality (participants affected / at risk) | 899/39750 | 866/39810
Serious Adverse Events (participants affected / at risk) | 0/39750 | 0/39810
Other Adverse Events (participants affected / at risk) | 0/39750 | 0/39810

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT03923699/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT03923699/SAP_001.pdf